CLINICAL TRIAL: NCT02149108
Title: A Double-blind, Randomised, Placebo Controlled Phase III Study of Nintedanib Plus Best Supportive Care (BSC) Versus Placebo Plus BSC in Patients With Metastatic Colorectal Cancer Refractory to Standard Therapies.
Brief Title: Nintedanib (BIBF 1120) vs Placebo in Refractory Metastatic Colorectal Cancer (LUME-Colon 1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1199.52; 2012-000095-42 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-06

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — nintedanib

ARMS (2):
- Nintedanib (BIBF 1120) + BSC (Experimental)
  Interventions: Drug: Nintedanib (BIBF 1120); Drug: BSC
- Placebo + BSC (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: BSC

INTERVENTIONS:
Drug: Nintedanib (BIBF 1120)
  Arms: Nintedanib (BIBF 1120) + BSC
Drug: Placebo
  Arms: Placebo + BSC
Drug: BSC
  Arms: Placebo + BSC
Drug: BSC
  Arms: Nintedanib (BIBF 1120) + BSC

SUMMARY:
The objective of this Phase III study is to evaluate the efficacy of nintedanib in patients with metastatic colorectal cancer (mCRC) after failure of previous treatment with standard chemotherapy and biological agents.

ELIGIBILITY:
Inclusion criteria:

* Age >= 18 years
* Signed informed consent
* Histologically or cytologically confirmed colorectal adenocarcinoma
* Metastatic or locally advanced disease not amenable to curative surgery and/or radiotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status = 1
* At least one measurable lesion according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1
* Progression on standard therapies or withdrawn from standard treatment due to unacceptable toxicity. Previous standard treatment must include all of the following:
* - fluoropyrimidine
* - oxaliplatin: Patients treated with oxaliplatin in adjuvant setting should have progressed within 6 months of completion of adjuvant therapy or they must have been treated with oxaliplatin for metastatic disease
* - irinotecan
* - bevacizumab or aflibercept
* - cetuximab or panitumumab for patients with K-Ras wt or Ras wt tumours
* - The remaining standard available therapy as recommended by investigator is best supportive care (note: previous treatment with regorafenib and TAS 102 are allowed and these agents should be administered before study if available to patient according to local standards)
* - Life expectancy of at least 12 weeks
* - Hepatic function: aspartate aminotransferase (AST)/ Alanine Amino Transferase (ALT) = 1.5 X Upper Limit of Normal (ULN) and bilirubin = ULN for patients without liver metastases. AST/ALT = 2.5 X ULN and bilirubin = ULN for patients with liver metastases. Patients with Gilbert syndrome and bilirubin < 2 X ULN and normal AST/ALT are eligible
* Coagulation parameters: International normalised ratio (INR) < 2 and partial prothrombin Time (PTT) = 2xULN

Exclusion criteria:

* Previous treatment with nintedanib
* toxicity attributed to previous anticancer therapy that did not resolve to Common Terminology Criteria for Adverse Events (CTCAE) grade =1
* History of other malignancies in the last 5 years, in particular those that could interfere with interpretation of results.
* Serious concomitant disease or medical condition affecting compliance with trial requirements or which are considered relevant for the evaluation of the efficacy or safety of the trial drug,
* Significant cardiovascular diseases
* History of severe haemorrhagic or thromboembolic event in the past 12 months
* Bleeding or thrombotic disorders requiring anticoagulant therapy such as warfarin, or similar agents requiring therapeutic INR monitoring
* Gastrointestinal disorders or abnormalities that would interfere with absorption of study drug
* Patient with brain metastases that are symptomatic and/or require therapy.
* Patients of childbearing potential who are sexually active and unwilling to use a highly effective method of contraception
* Pregnancy or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 768 (Actual)
Dates: Start 2014-09-25 (Actual); Primary Completion 2016-05-13 (Actual); Study Completion 2016-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (129):
- United States (14):
  - 1199.52.0108 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1199.52.0105 Boehringer Ingelheim Investigational Site, New Haven, Connecticut
  - 1199.52.0101 Boehringer Ingelheim Investigational Site, Plainville, Connecticut
  - 1199.52.0121 Boehringer Ingelheim Investigational Site, Arlington Heights, Illinois
  - 1199.52.0123 Boehringer Ingelheim Investigational Site, Sioux City, Iowa
  - 1199.52.0104 Boehringer Ingelheim Investigational Site, Topeka, Kansas
  - 1199.52.0114 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 1199.52.0113 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 1199.52.0125 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 1199.52.0119 Boehringer Ingelheim Investigational Site, Johnson City, New York
  - 1199.52.0115 Boehringer Ingelheim Investigational Site, Canton, Ohio
  - 1199.52.0106 Boehringer Ingelheim Investigational Site, Sylvania, Ohio
  - 1199.52.0102 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 1199.52.0120 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
- Argentina (5):
  - 1199.52.5404 Boehringer Ingelheim Investigational Site, Cdad. de Córdoba
  - 1199.52.5405 Boehringer Ingelheim Investigational Site, Cdad. de Córdoba
  - 1199.52.5401 Boehringer Ingelheim Investigational Site, Ciudad Autónoma de Bs As
  - 1199.52.5403 Boehringer Ingelheim Investigational Site, Ciudad Autónoma de Bs As
  - 1199.52.5406 Boehringer Ingelheim Investigational Site, Ciudad Autónoma de Bs As
- Australia (6):
  - 1199.52.6102 Boehringer Ingelheim Investigational Site, Concord, New South Wales
  - 1199.52.6103 Boehringer Ingelheim Investigational Site, St Leonards, New South Wales
  - 1199.52.6101 Boehringer Ingelheim Investigational Site, Wollongong, New South Wales
  - 1199.52.6104 Boehringer Ingelheim Investigational Site, Heidelberg, Victoria
  - 1199.52.6105 Boehringer Ingelheim Investigational Site, Nedlands, Western Australia
  - 1199.52.6106 Boehringer Ingelheim Investigational Site, Perth, Western Australia
- Austria (3):
  - 1199.52.4302 Boehringer Ingelheim Investigational Site, Linz
  - 1199.52.4303 Boehringer Ingelheim Investigational Site, Vienna
  - 1199.52.4304 Boehringer Ingelheim Investigational Site, Vienna
- Belgium (9):
  - 1199.52.3208 Boehringer Ingelheim Investigational Site, Aalst
  - 1199.52.3205 Boehringer Ingelheim Investigational Site, Bonheiden
  - 1199.52.3202 Boehringer Ingelheim Investigational Site, Brussels
  - 1199.52.3207 Boehringer Ingelheim Investigational Site, Charleroi
  - 1199.52.3204 Boehringer Ingelheim Investigational Site, Edegem
  - 1199.52.3203 Boehringer Ingelheim Investigational Site, Haine-Saint-Paul
  - 1199.52.3201 Boehringer Ingelheim Investigational Site, Leuven
  - 1199.52.3206 Boehringer Ingelheim Investigational Site, Liège
  - 1199.52.3521 Boehringer Ingelheim Investigational Site, Luxembourg
- Canada (4):
  - 1199.52.1003 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1199.52.1004 Boehringer Ingelheim Investigational Site, Edmonton, Ontario
  - 1199.52.1001 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1199.52.1002 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- Czechia (3):
  - 1199.52.4202 Boehringer Ingelheim Investigational Site, Brno
  - 1199.52.4204 Boehringer Ingelheim Investigational Site, Hradec Králové
  - 1199.52.4201 Boehringer Ingelheim Investigational Site, Prague
- Denmark (4):
  - 1199.52.4502 Boehringer Ingelheim Investigational Site, Herning
  - 1199.52.4501 Boehringer Ingelheim Investigational Site, København Ø
  - 1199.52.4503 Boehringer Ingelheim Investigational Site, Næstved
  - 1199.52.4504 Boehringer Ingelheim Investigational Site, Odense C
- France (4):
  - 1199.52.3304 Boehringer Ingelheim Investigational Site, Lille
  - 1199.52.3307 Boehringer Ingelheim Investigational Site, Lyon
  - 1199.52.3305 Boehringer Ingelheim Investigational Site, Paris
  - 1199.52.3301 Boehringer Ingelheim Investigational Site, Reims
- Germany (5):
  - 1199.52.4906 Boehringer Ingelheim Investigational Site, Dresden
  - 1199.52.4905 Boehringer Ingelheim Investigational Site, Essen
  - 1199.52.4904 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 1199.52.4903 Boehringer Ingelheim Investigational Site, Mannheim
  - 1199.52.4901 Boehringer Ingelheim Investigational Site, Ulm
- Hong Kong (4):
  - 1199.52.8501 Boehringer Ingelheim Investigational Site, Hong Kong
  - 1199.52.8502 Boehringer Ingelheim Investigational Site, Hong Kong
  - 1199.52.8503 Boehringer Ingelheim Investigational Site, Hong Kong
  - 1199.52.8504 Boehringer Ingelheim Investigational Site, Hong Kong
- Israel (3):
  - 1199.52.9706 Boehringer Ingelheim Investigational Site, Beersheba
  - 1199.52.9704 Boehringer Ingelheim Investigational Site, Petah Tikva
  - 1199.52.9703 Boehringer Ingelheim Investigational Site, Tel Aviv
- Italy (6):
  - 1199.52.3901 Boehringer Ingelheim Investigational Site, Genova
  - 1199.52.3906 Boehringer Ingelheim Investigational Site, Milan
  - 1199.52.3907 Boehringer Ingelheim Investigational Site, Napoli
  - 1199.52.3905 Boehringer Ingelheim Investigational Site, Padua
  - 1199.52.3903 Boehringer Ingelheim Investigational Site, Pisa
  - 1199.52.3904 Boehringer Ingelheim Investigational Site, San Giovanni Rotondo (FG)
- Japan (16):
  - 1199.52.8102 Boehringer Ingelheim Investigational Site, Aichi, Nagoya
  - 1199.52.8105 Boehringer Ingelheim Investigational Site, Chiba, Chiba
  - 1199.52.8101 Boehringer Ingelheim Investigational Site, Chiba, Kashiwa
  - 1199.52.8107 Boehringer Ingelheim Investigational Site, Ehime, Matsuyama
  - 1199.52.8106 Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - 1199.52.8108 Boehringer Ingelheim Investigational Site, Hokkaido, Sapporo
  - 1199.52.8115 Boehringer Ingelheim Investigational Site, Hyogo, Amagasaki
  - 1199.52.8112 Boehringer Ingelheim Investigational Site, Hyogo, Kobe
  - 1199.52.8114 Boehringer Ingelheim Investigational Site, Ibaraki, Tsukuba
  - 1199.52.8110 Boehringer Ingelheim Investigational Site, Oita, Yufu
  - 1199.52.8116 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1199.52.8103 Boehringer Ingelheim Investigational Site, Osaka, Suita
  - 1199.52.8109 Boehringer Ingelheim Investigational Site, Saitama, Kitaadachi-gun
  - 1199.52.8104 Boehringer Ingelheim Investigational Site, Shizuoka, Sunto-gun
  - 1199.52.8113 Boehringer Ingelheim Investigational Site, Tokyo , Shinagawa-ku
  - 1199.52.8111 Boehringer Ingelheim Investigational Site, Tokyo, Koto-ku
- 1199.52.5201 Boehringer Ingelheim Investigational Site, México, Mexico
- Netherlands (3):
  - 1199.52.3101 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1199.52.3103 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1199.52.3102 Boehringer Ingelheim Investigational Site, Utrecht
- Poland (3):
  - 1199.52.4801 Boehringer Ingelheim Investigational Site, Jelenia Góra
  - 1199.52.4803 Boehringer Ingelheim Investigational Site, Poznan
  - 1199.52.4804 Boehringer Ingelheim Investigational Site, Wroclaw
- Portugal (5):
  - 1199.52.3504 Boehringer Ingelheim Investigational Site, Almada
  - 1199.52.3502 Boehringer Ingelheim Investigational Site, Coimbra
  - 1199.52.3505 Boehringer Ingelheim Investigational Site, Loures
  - 1199.52.3501 Boehringer Ingelheim Investigational Site, Porto
  - 1199.52.3506 Boehringer Ingelheim Investigational Site, Porto
- Russia (4):
  - 1199.52.0701 Boehringer Ingelheim Investigational Site, Moscow
  - 1199.52.0703 Boehringer Ingelheim Investigational Site, Moscow
  - 1199.52.0702 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1199.52.0707 Boehringer Ingelheim Investigational Site, Tyumen
- South Korea (4):
  - 1199.52.8202 Boehringer Ingelheim Investigational Site, Goyang
  - 1199.52.8201 Boehringer Ingelheim Investigational Site, Seoul
  - 1199.52.8203 Boehringer Ingelheim Investigational Site, Seoul
  - 1199.52.8204 Boehringer Ingelheim Investigational Site, Seoul
- Spain (7):
  - 1199.52.3406 Boehringer Ingelheim Investigational Site, A Coruña
  - 1199.52.3401 Boehringer Ingelheim Investigational Site, Barcelona
  - 1199.52.3402 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat
  - 1199.52.3403 Boehringer Ingelheim Investigational Site, Madrid
  - 1199.52.3404 Boehringer Ingelheim Investigational Site, Madrid
  - 1199.52.3405 Boehringer Ingelheim Investigational Site, Santander
  - 1199.52.3407 Boehringer Ingelheim Investigational Site, Seville
- Sweden (2):
  - 1199.52.4601 Boehringer Ingelheim Investigational Site, Stockholm
  - 1199.52.4602 Boehringer Ingelheim Investigational Site, Uppsala
- Taiwan (4):
  - 1199.52.8805 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1199.52.8801 Boehringer Ingelheim Investigational Site, Taipei
  - 1199.52.8803 Boehringer Ingelheim Investigational Site, Taipei
  - 1199.52.8802 Boehringer Ingelheim Investigational Site, Taoyuan
- Turkey (Türkiye) (5):
  - 1199.52.9005 Boehringer Ingelheim Investigational Site, Adana
  - 1199.52.9001 Boehringer Ingelheim Investigational Site, Ankara
  - 1199.52.9003 Boehringer Ingelheim Investigational Site, Antalya
  - 1199.52.9004 Boehringer Ingelheim Investigational Site, Istanbul
  - 1199.52.9002 Boehringer Ingelheim Investigational Site, Izmir
- United Kingdom (5):
  - 1199.52.4401 Boehringer Ingelheim Investigational Site, Aberdeen
  - 1199.52.4403 Boehringer Ingelheim Investigational Site, Manchester
  - 1199.52.4402 Boehringer Ingelheim Investigational Site, Middlesex
  - 1199.52.4405 Boehringer Ingelheim Investigational Site, Nottingham
  - 1199.52.4404 Boehringer Ingelheim Investigational Site, Southampton

REFERENCES:
- [Derived] Van Cutsem E, Yoshino T, Lenz HJ, Lonardi S, Falcone A, Limon ML, Saunders M, Sobrero A, Park YS, Ferreiro R, Hong YS, Tomasek J, Taniguchi H, Ciardiello F, Stoehr J, Oum'Hamed Z, Vlassak S, Studeny M, Argiles G. Nintedanib for the treatment of patients with refractory metastatic colorectal cancer (LUME-Colon 1): a phase III, international, randomized, placebo-controlled study. Ann Oncol. 2018 Sep 1;29(9):1955-1963. doi: 10.1093/annonc/mdy241. PMID 30010751
- [Derived] Van Cutsem E, Yoshino T, Hocke J, Oum'Hamed Z, Studeny M, Tabernero J. Rationale and Design for the LUME-Colon 1 Study: A Randomized, Double-Blind, Placebo-Controlled Phase III Trial of Nintedanib Plus Best Supportive Care Versus Placebo Plus Best Supportive Care in Patients With Advanced Colorectal Cancer Refractory to Standard Treatment. Clin Colorectal Cancer. 2016 Mar;15(1):91-94.e1. doi: 10.1016/j.clcc.2015.09.005. Epub 2015 Oct 9. PMID 26603056

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The "completed" patients were on treatment (2 patients on Placebo, 3 patients on Nintedanib) at the data cut-off date 14JUN2016.
  The "NOT Completed" patients were off-treatment (380 patients on Placebo, 383 patients on Nintedanib) at the data cut-off date 14JUN2016.
Groups:
- Placebo: Placebo soft gelatin capsule matching that of Nintedanib twice daily (b.i.d.) administered orally of 21-day treatment course. If required the dose of placebo, could be reduced to 150 mg b.i.d. or 100 mg b.i.d. (according to the protocol-defined dose-reduction scheme). No dose increase was allowed after a dose reduction.
- Nintedanib: Nintedanib 200 mg twice daily (b.i.d.) administered orally in the form of a soft gelatin capsule of 21-day treatment course. If required the dose of Nintedanib, could be reduced to 150 mg b.i.d. or 100 mg b.i.d. (according to the protocol-defined dose-reduction scheme). No dose increase was allowed after a dose reduction.
Period: Overall Study
Arm/Group | Placebo | Nintedanib
Started | 382 (Randomised patients.) | 386 (Randomised patients.)
Completed | 2 (On-treatment at analysis cut-off date (14JUN2016).) | 3 (On-treatment at analysis cut-off date (14JUN2016).)
Not Completed | 380 | 383
Not completed — Not treated | 1 | 2
Not completed — Progressive Disease (PD) | 324 | 318
Not completed — Worsening/adverse event cancer disease | 31 | 32
Not completed — Other Adverse Event (AE) | 8 | 18
Not completed — Other not defined above | 0 | 2
Not completed — Refusal to continue trial medication | 15 | 11
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomised Set (RS): This patient set included all patients who were randomised to receive treatment, whether treated or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nintedanib | Total
Number analyzed (Participants) | 382 | 386 | 768
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.1 (10.8) | 61.0 (11.3) | 61.1 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164 | 150 | 314
  Male | 218 | 236 | 454

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) by Central Review Assessment
Description: PFS by central review assessment was defined as the time from the date of randomisation to the date of disease progression according to Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1 or death from any cause, whichever occurred first.
  Median, 95% Confidence Interval were calculated from an unadjusted Kaplan-Meier curve for each treatment arm.
Time Frame: From randomisation until cut-off date 14JUN2016.
Population: Randomised Set: This patient set included all patients who were randomised to receive treatment, whether treated or not.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Nintedanib
Number analyzed (Participants) | 382 | 386
Months | 1.38 [1.38 to 1.41] | 1.51 [1.45 to 2.17]
Statistical Analysis 1: Comparison: Placebo vs Nintedanib; Test type: Superiority or Other; p < 0.0001, Log Rank — Hazard ratio, confidence interval and p-value obtained from log-rank test stratified by regorafenib pre-treatment (yes vs no), time from onset metastatic disease until randomisation (less than 24 months vs 24 months or more ) and region; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.49 to 0.69] — Hazard ratio <1 favors Nintedanib

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomisation to the time of death from any cause.
  Median, 95% Confidence Interval were calculated from an unadjusted Kaplan-Meier curve for each treatment arm.
Time Frame: From randomisation until cut-off date 14JUN2016.
Population: Randomised Set: This patient set included all patients who were randomised to receive treatment, whether treated or not.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Nintedanib
Number analyzed (Participants) | 382 | 386
Months | 6.05 [5.22 to 6.97] | 6.44 [5.98 to 7.10]
Statistical Analysis 1: Comparison: Placebo vs Nintedanib; Test type: Superiority or Other; p = 0.8659, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.86 to 1.19] — Hazard ratio below 1 favors Nintedanib

3. Secondary Outcome: Objective Tumour Response (Complete Response (CR)) + Partial Response (PR) by Central Review Assessment
Description: Objective tumour response was defined as best overall response of CR or PR determined by central review assessment.
Time Frame: From randomisation until cut-off date 14JUN2016.
Population: Randomised Set: This patient set included all patients who were randomised to receive treatment, whether treated or not.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Nintedanib
Number analyzed (Participants) | 382 | 386
Percentage of participants | 0 | 0

4. Secondary Outcome: Disease Control (Complete Response + Partial Response + Stable Disease) by Central Review Assessment
Description: Disease control was defined as best overall response of CR, PR, or Stable Disease (SD).
Time Frame: From randomisation until cut-off date 14JUN2016.
Population: Randomised Set: This patient set included all patients who were randomised to receive treatment, whether treated or not.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Nintedanib
Number analyzed (Participants) | 382 | 386
Percentage of participants | 10.5 [3.68 to 6.67] | 25.6 [3.65 to 4.11]
Statistical Analysis 1: Comparison: Placebo vs Nintedanib; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Odds ratio and p-value are obtained from logistic regression model adjusted for regorafenib pre-treatment (yes vs no), time from onset metastatic disease until randomization in the trial (less than 24 months vs. 24 months or more) and region; Odds Ratio (OR) = 2.96, 95% CI 2-sided [2.00 to 4.47] — An odds ratio >1 indicates benefit to Nintedanib

ADVERSE EVENTS:
Time Frame: From first drug administration until 28 days after last drug administration, up to 22.7 months.
Description: 1. patient who was randomised to the Placebo was not treated. Consequently, number of subjects that started is 382 but only 381 reported that includes only treated patients.
  2. patients were randomised to the Nintedanib were not treated. Consequently, number of subjects that started is 386 but only 384 reported that includes only treated patients.
Arm/Group | Placebo | Nintedanib
Serious Adverse Events (participants affected / at risk) | 133/381 | 149/384
Other Adverse Events (participants affected / at risk) | 309/381 | 351/384
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=381) | Nintedanib (N=384)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 4 | 2
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 6
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 2
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1
Fistula of small intestine (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 2 | 5
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 6 | 6
Intestinal prolapse (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 3
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal obstruction (Gastrointestinal disorders) | 0 | 1
Rectal tenesmus (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 5
Asthenia (General disorders) | 3 | 4
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Condition aggravated (General disorders) | 1 | 0
Death (General disorders) | 4 | 2
Fatigue (General disorders) | 1 | 2
Gait disturbance (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 3 | 0
Generalised oedema (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 1 | 3
Performance status decreased (General disorders) | 3 | 5
Pyrexia (General disorders) | 4 | 3
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 4
Hepatic failure (Hepatobiliary disorders) | 4 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2
Jaundice (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 3
Oral candidiasis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 5 | 3
Postoperative wound infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 4
Septic shock (Infections and infestations) | 0 | 1
Small intestine gangrene (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 6
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 3 | 7
Aspartate aminotransferase increased (Investigations) | 5 | 6
Blood bilirubin increased (Investigations) | 6 | 2
Blood creatinine increased (Investigations) | 2 | 0
Hepatic enzyme increased (Investigations) | 0 | 2
Liver function test increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 5 | 6
Dehydration (Metabolism and nutrition disorders) | 1 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 24 | 27
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 3 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 2
Hemiparesis (Nervous system disorders) | 1 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 2
Paraparesis (Nervous system disorders) | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Sensory loss (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 7
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 5 | 4
Micturition disorder (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 3
Renal impairment (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 12
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0
Thrombosis in device (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=381) | Nintedanib (N=384)
Anaemia (Blood and lymphatic system disorders) | 22 | 23
Abdominal pain (Gastrointestinal disorders) | 59 | 65
Abdominal pain upper (Gastrointestinal disorders) | 21 | 25
Constipation (Gastrointestinal disorders) | 57 | 65
Diarrhoea (Gastrointestinal disorders) | 57 | 175
Nausea (Gastrointestinal disorders) | 103 | 163
Vomiting (Gastrointestinal disorders) | 71 | 149
Asthenia (General disorders) | 46 | 54
Fatigue (General disorders) | 89 | 113
Oedema peripheral (General disorders) | 28 | 22
Pain (General disorders) | 21 | 9
Pyrexia (General disorders) | 45 | 53
Alanine aminotransferase increased (Investigations) | 23 | 90
Aspartate aminotransferase increased (Investigations) | 44 | 90
Blood alkaline phosphatase increased (Investigations) | 22 | 28
Blood bilirubin increased (Investigations) | 15 | 26
Weight decreased (Investigations) | 13 | 35
Decreased appetite (Metabolism and nutrition disorders) | 96 | 128
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 30 | 33
Headache (Nervous system disorders) | 19 | 25
Insomnia (Psychiatric disorders) | 22 | 30
Proteinuria (Renal and urinary disorders) | 12 | 34
Cough (Respiratory, thoracic and mediastinal disorders) | 48 | 42
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40 | 35
Rash (Skin and subcutaneous tissue disorders) | 14 | 20
Hypertension (Vascular disorders) | 15 | 42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.